CLINICAL TRIAL: NCT02315911
Title: Randomized Controlled Studies of Sugery for Pediatric OSA: Part 1 Expectancy Compared to Adeno-tonsillectomy for Mild-moderate OSA. Part 2 Adeno-tonsillectomy Compared to Adeno-pharyngoplasty for Severe OSA.
Brief Title: Randomized Control Trials of Surgery for Pediatric OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Danielle Friberg, Ass professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCT02315911
Record Dates: First submitted 2014-12-08; First posted 2014-12-12 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Sleep Apnea, Obstructive; Otorhinolaryngologic Diseases; Pediatric Disorder
Keywords: Tonsillectomy; Adenoidectomy; Adenoidpharyngoplasty; OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive; Otorhinolaryngologic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- expectancy for mild-moderate OSA (No Intervention): 6 months expectancy
- ATE for mild-moderate OSA (Experimental): adeno-tonsillectomy
  Interventions: Procedure: ATE
- ATE for severe OSA (Experimental): adeno-tonsillectomy
  Interventions: Procedure: ATE
- APP for severe OSA (Experimental): adeno-pharyngoplasty
  Interventions: Procedure: APP

INTERVENTIONS:
Procedure: ATE — surgical removal of adenoids and tonsils
  Other Names: adeno-tonsillectomy
  Arms: ATE for mild-moderate OSA; ATE for severe OSA
Procedure: APP — surgical removal of adenoids and tonsils and suturing of palatal pillars
  Other Names: adeno-pharyngoplasty
  Arms: APP for severe OSA

SUMMARY:
Randomized study on pediatric OSA with 2 groups: mild-moderate OSA and severe OSA. Mild-moderate are randomized to either expectancy or ATE. Severe are randomized to either ATE or APP. Pediatric age span of 2 until 4,9 years.

DETAILED DESCRIPTION:
Children who are referred to ENT clinic because of sleep-disordered breathing and fulfil the inclusion criteria undergo polysomnography (PSG) and fill in questionnaires. Depending on the outcome of the PSG, whether a) the child have mild to moderate OSA (AHI between 2-9.9) the family is asked to be in the study. If yes, the doctor take a sealed envelope and open it, either the child are randomized to adenotonsillectomy (ATE) or 6 months expectancy. Whether PSG shows b) severe OSA and the family accept participation the child is operated within a month. There is a straification beetween 2 groups, if AHI is 1) between 10 and 29.9 or 2) above 30. A sealed envelope is open in the operating room by the surgeon. The child is randomized to either ATE or ATE and suturing of the tonsillar pillars. The study is blinded for the family, who will not know which method the child has undergone. After 6 months all children will undergo follow-up with PSG and questionnaires. If the expectancy group will deteriorate during waiting time, or the child still has moderate to severe OSA, they will undergo ATE. Further follow-ups at three and ten years. Altogether 160 children should be evaluated with two PSG, 80 in each group.

ELIGIBILITY:
Inclusion Criteria:

* OAHI >= 2
* Tonsillary hypertrophy, Brodsky size 2-4
* Adequate swedish knowledge

Exclusion Criteria:

* Cardiovascular disorders
* Pulmonary disorders
* Neuromuscular disorders
* Cranoifacial malformations
* Genetic disorders
* Earlier performed adenoid-tonsillary-surgery
* Bleeding disorders

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2014-12; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
obstructive apnea hypopnea index | 6 months
  with full-night polysomnography

SECONDARY OUTCOMES:
oxygen desaturation index | 6 months
  with full-night polysomnography
postoperative pain | 6 months
  visuell analog scale, questionnaire diaries. Number of days until normal diet.
per- and postoperative bleeding | postoperatively, weeks
  description of bleeding amount per and postoperatively, number of patients needed to reoperate because of bleeding postoperatively
quality of life | 6 months
  Questionnaires validated, SDQ and OSA-18
Innate lymphoid cells in tonsils | 6 months
  To investigate the amount of Innate lymphoid cells in children with OSA
side-effects of surgery | 6 months
  with a questionnaire evaluate if the child postoperatively will have speech-or swallowing difficulties. The parents will respond with a four-point Likert scale

OTHER OUTCOMES:
longterm results | 3 years
  with new polysomnography and questionnaires. Evaluate number of patients that are cured, AHI below 2.
longterm results | 10 years
  with new polysomnography and questionnaires.Evaluate number of patients that are cured, AHI below 2.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Tideholm, Study Director — ENT-clinic, Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Sjolander I, Fehrm J, Borgstrom A, Nerfeldt P, Friberg D. Adenotonsillectomy vs Watchful Waiting in Pediatric Mild to Moderate Obstructive Sleep Apnea: The KATE Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2025 Nov 1;151(11):1038-1045. doi: 10.1001/jamaoto.2025.2831. PMID 40965870
- [Derived] Fehrm J, Nerfeldt P, Browaldh N, Friberg D. Effectiveness of Adenotonsillectomy vs Watchful Waiting in Young Children With Mild to Moderate Obstructive Sleep Apnea: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2020 Jul 1;146(7):647-654. doi: 10.1001/jamaoto.2020.0869. PMID 32463430
- [Derived] Fehrm J, Nerfeldt P, Sundman J, Friberg D. Adenopharyngoplasty vs Adenotonsillectomy in Children With Severe Obstructive Sleep Apnea: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Jul 1;144(7):580-586. doi: 10.1001/jamaoto.2018.0487. PMID 29852045